CLINICAL TRIAL: NCT03519178
Title: PHASE 1/2A DOSE ESCALATION AND EXPANSION STUDY EVALUATING SAFETY, TOLERABILITY, PHARMACOKINETIC, PHARMACODYNAMICS AND ANTI-TUMOR ACTIVITY OF PF-06873600 AS A SINGLE AGENT AND IN COMBINATION WITH ENDOCRINE THERAPY
Brief Title: A Study of PF-06873600 in People With Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per business decision, but not due to safety concerns or regulatory request.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3661001; NCT03519178 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2018-02-22; First posted 2018-05-08 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: HR+ HER2- Metastatic Breast Cancer, Ovarian Cancer, Fallopian Tube Cancer, Primary Peritoneal Cancer, Triple Negative Breast Cancer, Male Breast Cancer
Keywords: Hormone Receptor (HR) Positive Breast Cancer; Estrogen receptor (ER) positive; Progesterone receptor (PR) positive; Cyclin-dependent kinase (CDK); Human epidermal growth factor receptor 2 (HER2) negative; Advanced breast cancer; Metastatic breast cancer (MBC); Triple negative breast cancer (TNBC); Epithelial ovarian cancer (EOC); Fallopian tube cancer; Primary peritoneal cancer (PPC); CDK4/6 inhibitor; Endocrine Therapy (ET); Measurable disease; Luteinizing Hormone Releasing Hormone (LHRH) Agonist; Goserelin; Leuprolide acetate
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms; Breast Neoplasms, Male; Breast Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation (Experimental): Single Agent Dose Escalation
  Interventions: Drug: PF-06873600
- Dose Finding Endocrine Therapy 1 Combination (Experimental): Part 1B PF-06873600 plus Endocrine Therapy 1
  Interventions: Drug: PF-06873600; Drug: Endocrine Therapy 1
- Dose Finding Endocrine Therapy 2 Combination (Experimental): Part 1B PF-06873600 plus Endocrine Therapy 2
  Interventions: Drug: PF-06873600; Drug: Endocrine Therapy 2
- Dose Expansion Arm A (Experimental): PF-06873600 as a Single Agent
  Interventions: Drug: PF-06873600
- Dose Expansion Arm B (Experimental): PF-06873600 as a Single Agent in Various Tumor Types
  Interventions: Drug: PF-06873600
- Dose Expansion Arm C (Experimental): PF-06873600 in Combination with Endocrine Therapy 1
  Interventions: Drug: PF-06873600; Drug: Endocrine Therapy 1
- Dose Expansion Arm D (Experimental): PF-06873600 in Combination with Endocrine Therapy 1
  Interventions: Drug: PF-06873600; Drug: Endocrine Therapy 1
- Dose Expansion Arm E (Experimental): PF-06873600 in Combination with Endocrine Therapy 2
  Interventions: Drug: PF-06873600; Drug: Endocrine Therapy 2

INTERVENTIONS:
Drug: PF-06873600 — PF-06873600 tablet for oral dosing
Drug: Endocrine Therapy 1 — Endocrine Therapy 1
  Arms: Dose Expansion Arm C; Dose Expansion Arm D; Dose Finding Endocrine Therapy 1 Combination
Drug: Endocrine Therapy 2 — Endocrine Therapy 2
  Arms: Dose Expansion Arm E; Dose Finding Endocrine Therapy 2 Combination

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of study medicine (PF-06873600) when taken alone or with hormone therapy by people with cancer.

People may be able to participate in this study if they have the following types of cancer: Hormone Receptor positive (HR+) breast cancer; Human Epidermal Growth Factor Receptor 2 (HER2)-negative breast cancer that is advanced or metastatic (spread to other parts of the body); triple negative breast cancer; epithelial ovarian cancer; fallopian tube cancer; or primary peritoneal cancer.

All participants in this study will receive the study medicine by mouth, 1 to 2 times a day at home. The dose of the study medicine may be changed during the study.

Some participants will also receive hormone therapy. The hormone therapy will be either letrozole by mouth once a day at home, or fulvestrant as a shot into the muscle. Fulvestrant will be given every two weeks at the study clinic for the first month, and then once a month after that.

Participants will take part in this study for at least 7 to 8 months, depending on how they respond to the therapy. During this time participants will visit the study clinic once a week for the first 2 cycles and every cycle thereafter.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, multi-center, non-randomized, multiple dose, safety, tolerability, pharmacokinetic, and pharmacodynamic study of PF-06873600 administered as a single agent in sequential dose levels and then in combination with endocrine therapy. In Part 1A and Part 1C, successive cohorts of patients will receive escalating doses of PF-06873600 and then in dose finding (Part 1B) with PF-06873600 in combination with endocrine therapy (ET). This study contains 2 parts, dose escalation with single agent (Part 1A and 1C) and then dose finding with PF-06873600 in combination with endocrine therapy (Part 1B) followed by dose expansion arms of PF-06873600 in combination with endocrine therapy (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) breast cancer

  • Prior combined CDK 4/6 inhibitor and endocrine therapy and 1 or 2 prior lines of chemotherapy
* Have a diagnosis of metastatic triple negative breast cancer (TNBC)

  • Up to 1-2 prior lines of chemotherapy
* Have a diagnosis of advanced platinum resistant epithelial ovarian cancer (EOC)/fallopian tube cancer/primary peritoneal cancer (PPC)

  • Up to 2-3 prior lines of therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Measurable disease or non-measurable disease and refractory to or intolerant of existing therapies (Part 1)
* Measurable disease as defined by RECIST 1.1 is required (Part 1B and Part 2 only)

Exclusion Criteria:

* Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases
* Other active malignancy within 3 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Major surgery or radiation within 4 weeks prior to study entry
* Last anti-cancer treatment within 2 weeks prior to study entry
* Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry
* Pregnant or breastfeeding female patients
* Active inflammatory gastrointestinal (GI) disease, known diverticular disease or previous gastric resection or lap band surgery including impairment of gastro intestinal function or GI disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University Of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center Pharmacy, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Highlands Oncology, Springdale, Arkansas
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Investigational Drugs Pharmacy, San Francisco, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - UCHealth Lone Tree Medical Center, Lone Tree, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute-Pharmacy, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - Rainier Hematology-Oncology PC, Puyallup, Washington
  - Rainier Hematology-Oncology, PC, Puyallup, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Bulgaria (3):
  - Multiprofile Hospital of Active Treatment - Dobrich AD, Dobrich
  - Specialized Hospital for Active Treatment of Oncology - Haskovo EOOD, Haskovo
  - Complex Oncology Center -Plovdiv, Plovdiv
- McGill University Health Centre, Montreal, Quebec, Canada
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa cancer center, Yokohama, Kanagawa
- Russia (4):
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - BIH of Omsk Region "Clinical Oncological Dispensary", Omsk
  - LLC "Medicina Severnoy Stolitsy", Saint Petersburg
  - LLC "Severo-Zapadny Medical Center", Saint Petersburg
- Ukraine (4):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, "Dnipro State Me, Dnipro, Dnipropetrovsk Oblast
  - Kharkiv Regional Specialized Dispensary of Radiation Protection of the Population, Kharkiv, Kharkivs’ka Oblast’
  - Communal nonprofit enterprise "Kyiv City Clinical Oncology Center" of Executive Body of Kyiv City, Kyiv
  - Communal noncommercial enterprise of Lviv regional council "Lviv oncological regional therapeutical, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3661001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) advanced or metastatic breast cancer (mBC), with locally recurrent/advanced or metastatic triple negative breast cancer (TNBC) or advanced platinum resistant ovarian/fallopian/peritoneal cancer, were recruited into this study. Two participants assigned to treatment but did not receive any study treatment were not included in any analysis.
Pre-assignment Details: Primary outcome measures and secondary outcome measures analysis was final at primary completion date milestone and reported on the same milestone.
Groups:
- Part 1A PF-06873600 1 mg Twice a Day (BID): Participants in Part 1A received PF-06873600 1 milligrams (mg) orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 2 mg BID: Participants in Part 1A received PF-06873600 2 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 5 mg BID: Participants in Part 1A received PF-06873600 5 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 10 mg BID: Participants in Part 1A received PF-06873600 10 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 25 mg BID: Participants in Part 1A received PF-06873600 25 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 25 mg BID Biomarker: Participants in Part 1A, with pre and on-treatment tumor and skin biopsies collected, received PF-06873600 25 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 35 mg BID: Participants in Part 1A received PF-06873600 35 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off: Participants in Part 1A received PF-06873600 35 mg orally intermittent dosing 5 days on/2 days off on a 28-day cycle, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1A PF-06873600 50 mg BID: Participants in Part 1A received PF-06873600 50 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination: Participants in Part 1B received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus fulvestrant 500 mg intramuscularly on Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2, and monthly thereafter, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or the study was terminated.
- Part 1B PF-06873600 25 mg BID IR/Letrozole Combination: Participants in Part 1B received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus letrozole 2.5 mg once daily as continuous daily dosing, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID: Participants in Part 1C received a single dose of PF-06873600 MR 20 mg orally during the lead-in period on Day -7 and Day -4, followed by IR 25 mg BID starting from Cycle 1 Day 1 orally BID on a 28-day cycle, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1C PF-06873600 MR 30 mg BID Long Release: Participants in Part 1C received PF-06873600 MR 30 mg BID starting from Cycle 1 Day 1 orally BID on a 28-day cycle, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination: Participants in Part 2A had received cyclin-dependent kinase 4/6 inhibitors (CDK4/6i) treatment before received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus fulvestrant 500 mg intramuscularly on Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2, and monthly thereafter, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination: Participants in Part 2C who were naïve to CDK4/6i received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus fulvestrant 500 mg intramuscularly on Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2, and monthly thereafter, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
Period: PF-06873600 Treatment
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Started | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 1
Not completed — Progressive disease | 1 | 1 | 1 | 1 | 6 | 7 | 3 | 7 | 3 | 5 | 4 | 3 | 4 | 28 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 3 | 2 | 0 | 2 | 1 | 1 | 2
Not completed — Global deterioration of health status | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 3 | 0
Not completed — Refused further treatment | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 9
Period: Fulvestrant. Treatment
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Started | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 9 | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 0 (This study period only applied to cohorts treated with fulvestrant.) | 45 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 45 | 28
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 30 | 8
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2
Not completed — Global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Period: Letrozole Treatment
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Started | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 7 | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.) | 0 (This study period only applied to cohorts treated with letrozole.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Follow-Up
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Started | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 0 (This study period did not apply to Part 2A.) | 0 (This study period did not apply to Part 2C.)
Completed | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 2 | 1 | 6 | 4 | 0 | 2 | 0 | 0
Not Completed | 1 | 2 | 2 | 3 | 5 | 4 | 3 | 11 | 9 | 3 | 3 | 5 | 4 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3 | 5 | 1 | 2 | 6 | 5 | 2 | 3 | 5 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-term Follow-up
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Started | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 0 (This study period only applied to Part 2.) | 45 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 28
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 19
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population consisted of all enrolled participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 Modified Release (MR) 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination | Total
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 1 | 7 | 6 | 3 | 11 | 7 | 6 | 6 | 2 | 4 | 34 | 17 | 108
  >=65 years | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 3 | 3 | 1 | 3 | 2 | 11 | 11 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28 | 151
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 12
  Not Hispanic or Latino | 1 | 2 | 2 | 3 | 8 | 6 | 2 | 10 | 9 | 7 | 6 | 4 | 6 | 37 | 27 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 5 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 10
  White | 1 | 2 | 1 | 3 | 4 | 6 | 3 | 8 | 8 | 9 | 4 | 5 | 2 | 32 | 20 | 108
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Part 1
Description: DLT was defined as any of the following adverse events (AEs) occurring in the first cycle of treatment (28 days) which were attributable to one, the other, or both agents in the combination: Hematologic - grade(G) 4 neutropenia lasting >7 days; Febrile neutropenia defined as an absolute neutrophil count (ANC) <1.0 * 10^9/L with a single temperature of >38.3°C, or a sustained temperature of ≥38°C, for more than 1 hour; G≥3 neutropenia with associated infection; G3 thrombocytopenia with clinically significant bleeding as indicated by ≥ G2 bleeding; G4 thrombocytopenia. Nonhematologic: Confirmed case of Drug Induced Liver Injury (DILI) (Hy's Law); G≥3 AEs that were clinically significant.
Time Frame: Cycle 1 (within 28 days after the first dose of study intervention)
Population: Analysis population consisted of all enrolled participants who received at least 1 dose of study intervention and who did not have major treatment deviations during the first cycle (ie, evaluable for the maximum tolerated dose [MTD]).
Measure: Count of Participants; unit: Participants
Groups:
- Part 1C PF-06873600 MR 20 IR 25 mg BID: Participants in Part 1C received a single dose of PF-06873600 MR 20 mg orally during the lead-in period on Day -7 and Day -4, followed by IR 25 mg BID starting from Cycle 1 Day 1 orally BID on a 28-day cycle
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 6 | 2 | 9 | 8 | 6 | 6 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) - Part 1 + Part 2
Description: An AE was defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occurred after participants' signed informed consent has been obtained. An SAE was an AE resulting in any of the following outcomes: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. Treatment Related AEs were treatment emergent AEs with cause categorized by the investigator as related to study treatment.
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 24 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Participants
  All-causality AEs | 1 | 2 | 2 | 3 | 9 | 6 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 25
  All-causality SAEs | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 4 | 6 | 1 | 2 | 0 | 3 | 9 | 5
  Treatment-related AEs | 0 | 2 | 1 | 0 | 8 | 6 | 4 | 13 | 10 | 8 | 7 | 5 | 5 | 45 | 24
  Treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 5 | 2

3. Primary Outcome: Number of Participants With Worst Post-Baseline Hematology Results Based on Common Terminology Criteria for Adverse Events (CTCAE) Grade: Part 1 + Part 2
Description: Severity was graded as NCI CTCAE version 4.03:Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 24 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study intervention. For each laboratory parameter, only participants with evaluable laboratory results were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 1 | 2 | 2 | 2 | 8 | 7 | 4 | 8 | 6 | 8 | 6 | 4 | 6 | 37 | 14
  Activated partial thromboplastin time prolonged: Grade 0 | 1 | 2 | 2 | 2 | 7 | 7 | 3 | 5 | 6 | 7 | 5 | 4 | 6 | 33 | 13
  Activated partial thromboplastin time prolonged: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 3 | 1
  Activated partial thromboplastin time prolonged: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Anemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Anemia: Grade 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 9 | 5
  Anemia: Grade 1 | 1 | 2 | 0 | 3 | 2 | 3 | 0 | 5 | 0 | 4 | 3 | 4 | 3 | 10 | 12
  Anemia: Grade 2 | 0 | 0 | 1 | 0 | 5 | 2 | 2 | 6 | 5 | 5 | 1 | 1 | 0 | 19 | 5
  Anemia: Grade 3 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 4 | 0 | 2 | 0 | 2 | 7 | 4
  Anemia: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Hemoglobin increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Hemoglobin increased: Grade 0 | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Hemoglobin increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  International normalized ratio (INR) increased: number analyzed (Participants) | 1 | 2 | 2 | 2 | 8 | 7 | 4 | 8 | 7 | 8 | 6 | 4 | 6 | 45 | 12
  International normalized ratio (INR) increased: Grade 0 | 1 | 2 | 2 | 2 | 7 | 7 | 3 | 8 | 6 | 7 | 6 | 4 | 6 | 29 | 9
  International normalized ratio (INR) increased: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 3
  International normalized ratio (INR) increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
  International normalized ratio (INR) increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  International normalized ratio (INR) increased: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Leukocytosis: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Leukocytosis: Grade 0 | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Leukocytosis: Grade 1 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Leukocytosis: Grade 2 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Leukocytosis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Lymphocyte count decreased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Lymphocyte count decreased: Grade 0 | 1 | 2 | 2 | 2 | 3 | 2 | 1 | 3 | 2 | 3 | 2 | 2 | 1 | 14 | 15
  Lymphocyte count decreased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 6 | 4
  Lymphocyte count decreased: Grade 2 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 6 | 1 | 1 | 4 | 0 | 4 | 21 | 5
  Lymphocyte count decreased: Grade 3 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 6 | 3 | 1 | 1 | 1 | 4 | 2
  Lymphocyte count decreased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Lymphocyte count increased: Grade 0 | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Lymphocyte count increased: Grade 1 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Lymphocyte count increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Neutrophil count decreased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Neutrophil count decreased: Grade 0 | 1 | 1 | 2 | 3 | 4 | 5 | 0 | 6 | 4 | 7 | 2 | 2 | 0 | 16 | 8
  Neutrophil count decreased: Grade 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 6 | 4
  Neutrophil count decreased: Grade 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 2 | 0 | 5 | 3 | 1 | 7 | 9
  Neutrophil count decreased: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 9 | 4
  Neutrophil count decreased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 7 | 1
  Platelet count decreased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  Platelet count decreased: Grade 0 | 1 | 2 | 2 | 3 | 6 | 5 | 0 | 9 | 5 | 5 | 4 | 3 | 4 | 28 | 17
  Platelet count decreased: Grade 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 14 | 8
  Platelet count decreased: Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Platelet count decreased: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Platelet count decreased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 26
  White blood cell decreased: Grade 0 | 1 | 1 | 2 | 1 | 4 | 2 | 0 | 0 | 3 | 2 | 0 | 2 | 0 | 11 | 7
  White blood cell decreased: Grade 1 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 7 | 0 | 4 | 1 | 1 | 1 | 8 | 7
  White blood cell decreased: Grade 2 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 5 | 3 | 3 | 6 | 2 | 4 | 16 | 8
  White blood cell decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 7 | 3
  White blood cell decreased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1

4. Primary Outcome: Number of Participants With Worst Post-Baseline Chemistry Results Based on Common Terminology Criteria for Adverse Events (CTCAE) Grade: Part 1 + Part 2
Description: as for outcome 3
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 24 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Participants
  Alanine aminotransferase increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Alanine aminotransferase increased: Grade 0 | 0 | 1 | 2 | 3 | 6 | 5 | 3 | 9 | 8 | 8 | 5 | 2 | 4 | 41 | 20
  Alanine aminotransferase increased: Grade 1 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 3 | 1 | 1 | 1 | 2 | 2 | 4 | 3
  Alanine aminotransferase increased: Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Alkaline phosphatase increased: Grade 0 | 1 | 1 | 2 | 2 | 5 | 5 | 2 | 9 | 6 | 6 | 4 | 2 | 1 | 31 | 16
  Alkaline phosphatase increased: Grade 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 4 | 3 | 3 | 2 | 4 | 13 | 6
  Alkaline phosphatase increased: Grade 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
  Alkaline phosphatase increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alkaline phosphatase increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Aspartate aminotransferase increased: Grade 0 | 0 | 1 | 2 | 2 | 5 | 6 | 2 | 9 | 7 | 6 | 3 | 2 | 2 | 38 | 16
  Aspartate aminotransferase increased: Grade 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 3 | 2 | 4 | 3 | 3 | 5 | 6
  Aspartate aminotransferase increased: Grade 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
  Aspartate aminotransferase increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Blood bilirubin increased: Grade 0 | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 8 | 9 | 7 | 5 | 6 | 45 | 19
  Blood bilirubin increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Blood bilirubin increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Creatinine increased: Grade 0 | 0 | 0 | 0 | 1 | 5 | 3 | 1 | 3 | 3 | 5 | 2 | 0 | 1 | 21 | 7
  Creatinine increased: Grade 1 | 1 | 2 | 2 | 2 | 4 | 4 | 3 | 8 | 5 | 4 | 5 | 5 | 5 | 22 | 17
  Creatinine increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0
  Creatinine increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypercalcemia: Grade 0 | 1 | 2 | 2 | 3 | 7 | 4 | 4 | 12 | 8 | 7 | 7 | 3 | 5 | 38 | 22
  Hypercalcemia: Grade 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 5 | 2
  Hypercalcemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Hypercalcemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperglycemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hyperglycemia: Grade 0 | 1 | 2 | 2 | 2 | 6 | 5 | 4 | 10 | 6 | 6 | 5 | 5 | 4 | 23 | 12
  Hyperglycemia: Grade 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 4 | 3 | 1 | 0 | 2 | 18 | 8
  Hyperglycemia: Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Hyperglycemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
  Hyperglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hyperkalemia: Grade 0 | 0 | 2 | 2 | 3 | 8 | 7 | 4 | 12 | 9 | 9 | 7 | 5 | 4 | 42 | 23
  Hyperkalemia: Grade 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Hyperkalemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypermagnesemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypermagnesemia: Grade 0 | 1 | 2 | 1 | 3 | 9 | 7 | 4 | 12 | 7 | 9 | 6 | 5 | 6 | 42 | 15
  Hypermagnesemia: Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 3 | 8
  Hypermagnesemia: Grade 2 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Hypermagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypermagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypernatremia: Grade 0 | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 8 | 9 | 7 | 5 | 6 | 44 | 24
  Hypernatremia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypoalbuminemia: Grade 0 | 1 | 2 | 2 | 2 | 4 | 4 | 3 | 11 | 5 | 8 | 6 | 5 | 5 | 35 | 18
  Hypoalbuminemia: Grade 1 | 0 | 0 | 0 | 1 | 5 | 3 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 7 | 5
  Hypoalbuminemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1
  Hypoalbuminemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Hypocalcemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypocalcemia: Grade 0 | 1 | 2 | 2 | 3 | 8 | 7 | 4 | 10 | 7 | 7 | 4 | 5 | 6 | 36 | 13
  Hypocalcemia: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 3 | 0 | 0 | 7 | 9
  Hypocalcemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Hypocalcemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypocalcemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypoglycemia: Grade 0 | 1 | 2 | 2 | 3 | 8 | 7 | 3 | 13 | 10 | 8 | 7 | 5 | 6 | 44 | 23
  Hypoglycemia: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Hypoglycemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypokalemia: Grade 0 | 1 | 2 | 2 | 2 | 8 | 6 | 3 | 10 | 7 | 8 | 6 | 5 | 5 | 33 | 19
  Hypokalemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 11 | 4
  Hypokalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
  Hypokalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypomagnesemia: Grade 0 | 1 | 2 | 2 | 1 | 5 | 4 | 3 | 7 | 8 | 3 | 2 | 5 | 4 | 24 | 14
  Hypomagnesemia: Grade 1 | 0 | 0 | 0 | 2 | 4 | 2 | 1 | 5 | 2 | 6 | 5 | 0 | 2 | 20 | 10
  Hypomagnesemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypomagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hyponatremia: Grade 0 | 1 | 1 | 0 | 1 | 5 | 3 | 3 | 12 | 3 | 8 | 5 | 4 | 3 | 40 | 20
  Hyponatremia: Grade 1 | 0 | 1 | 2 | 2 | 4 | 4 | 1 | 1 | 7 | 1 | 2 | 1 | 3 | 5 | 3
  Hyponatremia: Grade 2 | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03. | NA — Not defined in CTCAE v4.03.
  Hyponatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyponatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Hypophosphatemia: Grade 0 | 1 | 2 | 2 | 3 | 7 | 5 | 3 | 9 | 8 | 7 | 6 | 5 | 6 | 39 | 22
  Hypophosphatemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Hypophosphatemia: Grade 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 3 | 0
  Hypophosphatemia: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypophosphatemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Lipase increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Lipase increased: Grade 0 | 1 | 1 | 2 | 3 | 9 | 6 | 4 | 11 | 9 | 7 | 6 | 5 | 5 | 42 | 15
  Lipase increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 5
  Lipase increased: Grade 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Lipase increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Lipase increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Serum amylase increased: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 24
  Serum amylase increased: Grade 0 | 1 | 2 | 2 | 3 | 9 | 6 | 4 | 12 | 9 | 7 | 5 | 5 | 6 | 41 | 20
  Serum amylase increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 3 | 4
  Serum amylase increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Serum amylase increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Serum amylase increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Post-Baseline Vital Sign Abnormalities Meeting Pre-Defined Categorization - Part 1 + Part 2
Description: Pre-defined criteria included: 1) systolic blood pressure (SBP) (mm Hg) minimum (min) value <90; 2) SBP change from baseline (CFB) (mm Hg) maximum (max) decrease >=30 or max increase >=30; 3) diastolic blood pressure (DBP) (mm Hg) min <50; 4) DBP CFB (mm Hg) max decrease >=20 or max increase >=20; 5) supine heart rate (HR) beats per minute (bpm) min <40 or max >120.
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 24 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study intervention. For each vital sign measurement, only participants with evaluable vital sign results were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Participants
  SBP (mm Hg) <90: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  SBP (mm Hg) <90 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0
  SBP CFB (mm Hg) >= 30 increase: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  SBP CFB (mm Hg) >= 30 increase | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 5 | 2
  SBP CFB (mm Hg) >= 30 decrease: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  SBP CFB (mm Hg) >= 30 decrease | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 0 | 13 | 2
  DBP (mm Hg) <50: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  DBP (mm Hg) <50 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
  DBP CFB (mm Hg) >=20 increase: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  DBP CFB (mm Hg) >=20 increase | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 2 | 4
  DBP CFB (mm Hg) >=20 decrease: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  DBP CFB (mm Hg) >=20 decrease | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 10 | 4
  Heart rate (bpm) <40: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  Heart rate (bpm) <40 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Heart rate (bpm) >120: number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 27
  Heart rate (bpm) >120 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Changes Meeting Pre-Defined Categorization - Part 1 + Part 2
Description: ECG pre-defined categories for QTc interval adjusted according to Fridericia formula (QTcF) (msec) included: 450 <= max. <=480, 481 <= max. <=500, max >=501; QTcF CFB: 30 < max <=60, max >60; for PR and QRS: PR (msec): max >=300; PR increase from baseline: Baseline >200 and max. >=25% increase, Baseline <=200 and max. >=50% increase; QRS (msec): max >=200; QRS (msec) increase from baseline: Baseline >100 and max. >=25% increase, Baseline <=100 and max. >=50% increase. Categories, with at least 1 participant having ECG abnormality in any of the reporting arms, were reported in this outcome measure.
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 24 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study intervention. Only participants with evaluable ECG results were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 7 | 5 | 6 | 45 | 28
Participants
  PR interval not otherwise specified (NOS) (msec) baseline >200 and percent change >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PR interval NOS (msec) baseline <=200 and percent change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  QRS interval not otherwise specified (NOS) (msec): baseline >100 and change from baseline >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QRS interval not otherwise specified (NOS) (msec): baseline <=100 and change from baseline >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF NOS (msec): 450 <= value <=480 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 6 | 1 | 3 | 4 | 3 | 2 | 14 | 5
  QTcF NOS (msec): 481 <= value <=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  QTcF NOS (msec): value >=501 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  QTcF NOS (msec): 30 <= change from baseline <=60 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 9 | 5
  QTcF NOS (msec): change from baseline >60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2

7. Primary Outcome: Overall Response Rate (ORR): Part 2
Description: ORR: percentage of participants with confirmed complete response (CR) or partial response (PR). Response evaluation criteria in solid tumors (RECIST) v1.1: a) CR = disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions that had a reduction in short axis to less than (<) 10 millimeter (mm). Disappearance of all non-target lesions. In addition, all lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis) and b) PR = at least a 30 percent (%) decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Any radiological assessments taken more than 30 days after the last dose of study therapy or after antineoplastic agents other than study treatments taken by the participants was excluded from the best overall response derivation. Confirmation of CR or PR was to be at least 4 weeks apart from the previous radiological assessment.
Time Frame: From the start of the treatment until disease/clinical progression or death or early study discontinuation, whichever happened earlier (approximately up to 24 months)
Population: For Part 2: the response evaluable population included all participants who received at least 1 dose of study treatment and had baseline disease and at least 1 post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 45 | 22
Percentage of participants | 6.7 [1.4 to 18.3] | 22.7 [7.8 to 45.4]

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1 + Part 2
Description: The maximum observed concentration of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B and Part 2) was reported. The Cmax value was observed directly from data.
Time Frame: Part 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on Cycle 1 Day 1 (C1D1); Part 2: pre-dose, 1, 2, 4, 6 hours post-dose on C1D1
Population: The PK parameter analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Geometric Coefficient of Variation was not presented for parameters with participants with evaluable data <3 at that time point. For groups where 2 participants were evaluable for the PK parameter, exact data were presented, instead of the geometric mean (geometric coefficient of variation [CV]).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 6 | 5 | 6 | 43 | 24
Nanogram per milliliter | 5.39 (NA) — Only 1 participant evaluable. | 22.1 (31.9) | 29.1 (90.8) | 164.1 (37) | 243.5 (47) | 202.6 (47) | 388.1 (9) | 276.4 (42) | 393.8 (42) | 225.4 (28) | 228.5 (32) | 121.8 (54) | 43.51 (121) | 224.9 (43) | 181.4 (41)

9. Secondary Outcome: Time to Reach Cmax at Steady State (Tmax) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1 + Part 2
Description: Tmax of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B and Part 2) was reported.
Time Frame: Part 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1; Part 2: pre-dose, 1, 2, 4, 6 hours post-dose on C1D1
Population: The PK parameter analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 6 | 5 | 6 | 43 | 24
Hour | 2.17 [2.17 to 2.17] | 1.25 [0.500 to 2.00] | 2.02 [2.00 to 2.03] | 0.983 [0.500 to 1.90] | 2.17 [1.10 to 5.47] | 1.90 [0.517 to 3.00] | 3.64 [2.00 to 5.92] | 2.02 [0.517 to 6.00] | 3.49 [0.550 to 6.03] | 1.97 [0.533 to 5.95] | 2.52 [0.500 to 3.00] | 2.00 [0.517 to 10.3] | 10.0 [5.35 to 10.2] | 1.98 [1.00 to 4.17] | 1.94 [0.967 to 5.50]

10. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1
Description: AUClast of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1
Population: The PK parameter analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Geometric Coefficient of Variation was not presented for parameters with participants with evaluable data <3 at that time point. For groups where 2 participants were evaluable for the PK parameter, exact data were presented, instead of the geometric mean (geometric CV).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 4 | 13 | 10 | 9 | 6 | 5 | 6
Hour*nanogram per milliliter | 18.3 (NA) — Only 1 participant evaluable. | 39.2 (58.3) | 96.6 (442) | 599.4 (53) | 1295 (25) | 787.9 (59) | 2510 (25) | 1395 (38) | 1976 (49) | 1034 (43) | 1040 (46) | 596.8 (33) | 192.0 (201)

11. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1
Description: AUCinf of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 6 | 5 | 2 | 9 | 4 | 6 | 6 | 5 | 0
Hour*nanogram per milliliter | 21.0 (NA) — Only 1 participant evaluable. | 45.2 (NA) — Only 1 participant evaluable. | 101 (NA) — Only 1 participant evaluable. | 648.4 (60) | 1492 (20) | 892.6 (73) | 2010 (3400) | 1614 (48) | 1875 (41) | 884.3 (34) | 1142 (50) | 593.3 (17) |

12. Secondary Outcome: Apparent Clearance (CL/F) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1
Description: CL/F of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 6 | 5 | 2 | 9 | 4 | 6 | 6 | 3 | 0
Liter per hour | 47.6 (NA) — Only 1 participant evaluable. | 44.2 (NA) — Only 1 participant evaluable. | 49.7 (NA) — Only 1 participant evaluable. | 15.43 (60) | 16.78 (20) | 28.04 (73) | 10.3 (17.4) | 21.70 (48) | 26.63 (41) | 28.26 (34) | 21.87 (50) | 42.14 (17) |

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1
Description: Vz/F of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 6 | 5 | 2 | 9 | 4 | 6 | 6 | 3 | 0
Liter | 111 (NA) — Only 1 participant evaluable. | 116 (NA) — Only 1 participant evaluable. | 141 (NA) — Only 1 participant evaluable. | 55.32 (28) | 61.33 (20) | 97.32 (56) | 55.5 (60.0) | 86.06 (37) | 79.74 (15) | 83.54 (17) | 72.18 (37) | 132.2 (52) |

14. Secondary Outcome: Terminal Half-life (t1/2) of PF-06873600 Following a Single Oral Dose of Study Intervention on Cycle 1 Day 1 - Part 1
Description: t1/2 of PF-06873600 after single dose of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D1
Population: The PK parameter analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Standard deviation was not presented for parameters with participants with evaluable data <3 at that time point. For groups where 2 participants were evaluable for the PK parameter, exact data were presented, instead of the mean (standard deviation).
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 6 | 5 | 2 | 9 | 4 | 6 | 6 | 3 | 0
Hour | 1.61 (NA) — Only 1 participant evaluable. | 1.82 (NA) — Only 1 participant evaluable. | 1.96 (NA) — Only 1 participant evaluable. | 2.567 (0.82033) | 2.540 (0.14394) | 2.446 (0.54574) | 2.39 (3.74) | 2.809 (0.59669) | 2.163 (0.74732) | 2.128 (0.73966) | 2.428 (0.87316) | 2.250 (0.77350) |

15. Secondary Outcome: Steady State Maximum Concentration (Css,Max) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1 + Part 2
Description: Css,max of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B and Part 2) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: Part 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D15; Part 2: pre-dose, 1, 2, 4, 6 hours post-dose on C1D15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 2 | 9 | 6 | 8 | 7 | 6 | 39 | 21
Nanogram per milliliter | 10.9 (NA) — Only 1 participant evaluable. | 18.2 (45.4) | 46.3 (126) | 124.3 (29) | 382.4 (33) | 246.4 (40) | 362 (399) | 290.2 (29) | 335.2 (22) | 305.0 (35) | 276.5 (31) | 82.11 (72) | 273.5 (35) | 250.5 (44)

16. Secondary Outcome: Time to Maximum Plasma Concentration at Steady State (Tss,Max) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1 + Part 2
Description: Tss,max of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B and Part 2) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 2 | 9 | 6 | 8 | 7 | 6 | 39 | 21
Hour | 1.00 [1.00 to 1.00] | 1.25 [0.500 to 2.00] | 1.20 [0.500 to 1.90] | 2.00 [0.250 to 2.13] | 1.95 [0.900 to 5.70] | 1.92 [1.00 to 2.92] | 2.01 [2.00 to 2.02] | 2.23 [0.000 to 4.05] | 1.98 [1.10 to 4.25] | 1.88 [0.517 to 2.12] | 2.08 [1.82 to 3.93] | 2.99 [0.000 to 4.00] | 1.95 [0.917 to 4.02] | 1.97 [0.933 to 5.88]

17. Secondary Outcome: Steady State Minimum Plasma Concentration (Css,Min) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1 + Part 2
Description: Css,min of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B and Part 2) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 2 | 9 | 6 | 8 | 7 | 6 | 38 | 21
Nanogram per milliliter | 0.0000 (NA) — Only 1 participant evaluable. | 0.000 (0.000) | 1.19 (23.6) | 5.499 (5) | 37.63 (112) | 21.28 (130) | 52.1 (80.4) | 25.56 (8) | 25.63 (101) | 21.25 (106) | 13.33 (204) | 45.78 (49) | 23.67 (156) | 19.16 (131)

18. Secondary Outcome: Steady-State Area Under the Plasma Concentration Versus Time Curve Within One Dose Interval (AUCss,Tau) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1
Description: AUCss,tau of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 2 | 7 | 4 | 8 | 7 | 6
Hour*nanogram per milliliter | 25.3 (NA) — Only 1 participant evaluable. | 51.4 (86.9) | 150 (483) | 448.8 (25) | 1695 (34) | 1010 (40) | 2060 (2360) | 1372 (39) | 1607 (34) | 1229 (41) | 1273 (50) | 636.8 (59)

19. Secondary Outcome: Steady-State Apparent Oral Plasma Clearance (CLss/F) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1
Description: CLss/F of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 9 | 7 | 2 | 7 | 4 | 7 | 7 | 6
Liter per hour | 39.5 (NA) — Only 1 participant evaluable. | 23.0 (38.9) | 10.4 (33.2) | 22.28 (24) | 14.78 (34) | 24.76 (40) | 14.8 (17.0) | 25.54 (39) | 21.99 (44) | 20.35 (41) | 19.63 (49) | 47.08 (59)

20. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1
Description: Vss/F of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 0 | 2 | 1 | 3 | 6 | 6 | 1 | 6 | 4 | 6 | 5 | 0
Liter |  | 53.3 (98.4) | 124 (NA) — Only 1 participant evaluable. | 72.17 (19) | 57.62 (29) | 99.62 (35) | 70.8 (NA) — Only 1 participant evaluable. | 99.03 (48) | 75.41 (17) | 75.71 (32) | 80.33 (27) |

21. Secondary Outcome: Accumulation Ratio Based on AUC (Rac) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 1
Description: Rac of PF-06873600 after multiple doses of study intervention when given as a single agent (Part 1A and Part 1C), in combination with letrozole, and in combination with fulvestrant (Part 1B) was reported. Multiple-dose PK parameters were not calculated for the modified release selection cohort in Part 1C (ie, the group "Part 1C PF-06873600 MR 20 IR 25 mg BID").
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 12 hours post-dose on C1D15
Population: The PK parameter analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Geometric Coefficient of Variation was not presented for parameters with participants with evaluable data <3 at that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID Immediate Release (IR)/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 30 mg BID Long Release
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 6 | 5 | 1 | 5 | 4 | 5 | 6 | 0
Ratio | 1.210 (NA) — Only 1 participant evaluable. | 1.160 (NA) — Only 1 participant evaluable. | 1.53 (NA) — Only 1 participant evaluable. | 0.7263 (28) | 1.045 (17) | 1.254 (49) | 0.822 (NA) — Only 1 participant evaluable. | 0.8893 (32) | 1.260 (25) | 1.191 (29) | 1.268 (35) |

22. Secondary Outcome: Accumulation Ratio Based on Cmax (Observed) (Rac,Cmax) of PF-06873600 Following Multiple Doses of Study Intervention on Cycle 1 Day 15 - Part 2
Description: Rac,cmax of PF-06873600 after multiple doses of study intervention when given as in combination with fulvestrant (Part 2) was reported.
Time Frame: Pre-dose, 1, 2, 4, 6 hours post-dose on C1D15
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 36 | 19
Ratio | 1.161 (78) | 1.381 (34)

23. Secondary Outcome: Pharmacodynamic (PD) Biomarker Phospho-retinoblastoma Protein (pRb) in Tumor Tissue in Participants - Part 1 + Part 2
Description: Level of the PD marker, pRb, was analyzed at 2 time points, at screening and at Cycle 2 Day 1. Percentage changes of pRb at Cycle 2 Day 1 from screening (baseline) were calculated.
Time Frame: Screening and Cycle 2 Day 1
Population: The biomarker analysis population was all enrolled participants with PD biomarkers evaluated at pre-and/post dose.
Measure: Median (95% Confidence Interval); unit: Percentage of change
Groups:
- Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination: Participants in Part 1B received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus fulvestrant 500 mg intramuscularly on Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2, and monthly thereafter, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or the study was terminated.
Arm/Group | Part 1A PF-06873600 1 mg Twice a Day (BID) | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 0
Percentage of change |  |  |  |  | -84.44 [NA to NA] — Only 1 participant evaluable. | -11.11 [-172.414 to 326.323] |  |  |  |  | -77.50 [NA to NA] — Only 1 participant evaluable. |  |  | -30.43 [-103.371 to 184.820] |

24. Secondary Outcome: PD Biomarker Ki67 in Tumor Tissue in Participants - Part 1 + Part 2
Description: Level of the PD marker, Ki67, was analyzed at 2 time points, at screening and at Cycle 2 Day 1. Percent changes of pRb at Cycle 2 Day 1 from screening (baseline) were calculated.
Time Frame: Screening and Cycle 2 Day 1
Population: The biomarker analysis population was all enrolled participants with PD biomarkers evaluated at pre-and/post dose.
Measure: Median (95% Confidence Interval); unit: Percentage of change
Groups:
- Part 1A PF-06873600 1 mg BID: Participants in Part 1A received PF-06873600 1 milligrams (mg) orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
Arm/Group | Part 1A PF-06873600 1 mg BID | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 0
Percentage of change |  |  |  |  | -63.64 [NA to NA] — Only 1 participant evaluable. | -6.67 [-99.910 to 138.742] |  |  |  |  | -90.00 [NA to NA] — Only 1 participant evaluable. |  |  | -33.33 [-60.398 to 8.593] |

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after the last dose of study intervention, up to approximately 36.6 months
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or one participant may have experienced both a serious and non-serious event during the study. The safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Groups:
- Part 1A PF-06873600 1 mg BID: Participants in Part 1A received PF-06873600 1 mg orally BID on a 28-day cycle from Day 1 to Day 28, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 1C PF-06873600 MR 20 mg IR 25 mg BID: Participants in Part 1C received a single dose of PF-06873600 MR 20 mg orally during the lead-in period on Day -7 and Day -4, followed by IR 25 mg BID starting from Cycle 1 Day 1 orally BID on a 28-day cycle, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
- Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination: Participants in Part 2A had received CDK4/6i treatment before received PF-06873600 IR 25 mg orally BID on a 28-day cycle from Day 1 to Day 28 plus fulvestrant 500 mg intramuscularly on Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2, and monthly thereafter, until progression of disease, uncontrollable toxicity, a decision by the participant or investigator to discontinue treatment, or study termination.
Arm/Group | Part 1A PF-06873600 1 mg BID | Part 1A PF-06873600 2 mg BID | Part 1A PF-06873600 5 mg BID | Part 1A PF-06873600 10 mg BID | Part 1A PF-06873600 25 mg BID | Part 1A PF-06873600 25 mg BID Biomarker | Part 1A PF-06873600 35 mg BID | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off | Part 1A PF-06873600 50 mg BID | Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination | Part 1C PF-06873600 MR 20 mg IR 25 mg BID | Part 1C PF-06873600 MR 30 mg BID Long Release | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/2 | 0/3 | 1/9 | 0/7 | 0/4 | 1/13 | 3/10 | 1/9 | 0/7 | 0/5 | 3/6 | 6/45 | 4/28
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/2 | 0/3 | 2/9 | 0/7 | 1/4 | 4/13 | 6/10 | 1/9 | 2/7 | 0/5 | 3/6 | 9/45 | 5/28
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 2/2 | 3/3 | 9/9 | 6/7 | 4/4 | 13/13 | 10/10 | 9/9 | 7/7 | 5/5 | 6/6 | 45/45 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-06873600 1 mg BID (N=1) | Part 1A PF-06873600 2 mg BID (N=2) | Part 1A PF-06873600 5 mg BID (N=2) | Part 1A PF-06873600 10 mg BID (N=3) | Part 1A PF-06873600 25 mg BID (N=9) | Part 1A PF-06873600 25 mg BID Biomarker (N=7) | Part 1A PF-06873600 35 mg BID (N=4) | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off (N=13) | Part 1A PF-06873600 50 mg BID (N=10) | Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination (N=9) | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination (N=7) | Part 1C PF-06873600 MR 20 mg IR 25 mg BID (N=5) | Part 1C PF-06873600 MR 30 mg BID Long Release (N=6) | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination (N=45) | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-06873600 1 mg BID (N=1) | Part 1A PF-06873600 2 mg BID (N=2) | Part 1A PF-06873600 5 mg BID (N=2) | Part 1A PF-06873600 10 mg BID (N=3) | Part 1A PF-06873600 25 mg BID (N=9) | Part 1A PF-06873600 25 mg BID Biomarker (N=7) | Part 1A PF-06873600 35 mg BID (N=4) | Part 1A PF-06873600 35 mg Intermittent Dosing 5 Days on / 2 Days Off (N=13) | Part 1A PF-06873600 50 mg BID (N=10) | Part 1B PF-06873600 25 mg BID IR/Fulvestrant Combination (N=9) | Part 1B PF-06873600 25 mg BID IR/Letrozole Combination (N=7) | Part 1C PF-06873600 MR 20 mg IR 25 mg BID (N=5) | Part 1C PF-06873600 MR 30 mg BID Long Release (N=6) | Part 2A PF-06873600 25 mg BID IR/Fulvestrant Combination (N=45) | Part 2C PF-06873600 25 mg BID IR/Fulvestrant Combination (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 4 | 4 | 6 | 5 | 5 | 3 | 3 | 21 | 11
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 10 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 4 | 4 | 1 | 2 | 4 | 13 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 4 | 1 | 3 | 1 | 0 | 13 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 6 | 5 | 0 | 9 | 6 | 6 | 5 | 2 | 4 | 30 | 20
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 5 | 6 | 2 | 3 | 1 | 1 | 17 | 13
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 8 | 3 | 3 | 3 | 0 | 1 | 28 | 6
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 3
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 4 | 3
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 4 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 2 | 2 | 2 | 5 | 3 | 4 | 18 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 1 | 1 | 4 | 1 | 2 | 1 | 6 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 3 | 4 | 1 | 3 | 9 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 8 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 4 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 2 | 1 | 0 | 0 | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 12 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 4
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4 | 3 | 1 | 1 | 2 | 1 | 18 | 10
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 4 | 0 | 0 | 0 | 1 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 2 | 4 | 1 | 2 | 2 | 0 | 17 | 8
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03519178/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03519178/SAP_001.pdf